CLINICAL TRIAL: NCT07229872
Title: A Phase II Clinical Study of Aipalolitovorelizumab (QL1706) Combined With Fruquintinib in the Treatment of Immunodominant pMMR/MSS Metastatic Colorectal Cancer That Has Failed Second-line or Above Treatment
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Harbin Medical University (Other)
Responsible Party: Principal Investigator, Yanqiao Zhang, professor, Harbin Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QL-CRC-QIBA-3007
Record Dates: First submitted 2025-08-05; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Immunotherapy; Microsatellite stability; Immune advantage
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm experimental group (Experimental): Participants will receive:
  Aipalolitovorelizumab (QL1706) injection at a dose of 5mg/kg, administered intravenously on Day 1 of each 3-week treatment cycle.
  Fruquintinib at a dose of 5mg per day, taken orally continuously for the first 2 weeks of each 3-week cycle, followed by 1 week of withdrawal.
  Interventions: Drug: Aipalolitovorelizumab; Drug: Fruquintinib

INTERVENTIONS:
Drug: Aipalolitovorelizumab — Aipalolitovorelizumab (QL1706) injection at a dose of 5mg/kg, administered intravenously on Day 1 of each 3-week treatment cycle.
Drug: Fruquintinib — Fruquintinib at a dose of 5mg per day, taken orally continuously for the first 2 weeks of each 3-week cycle, followed by 1 week of withdrawal.

SUMMARY:
The goal of this clinical trial is to explore the preliminary efficacy and tolerability of Aipalolitovorelizumab (QL1706) in combination with fruquintinib for the treatment of metastatic colorectal cancer patients with immunodominant pMMR/MSS type who have failed second-line or above treatment. It is an open-label, single-arm, single-center phase II trial. The main questions it aims to answer are:

What is the objective response rate (ORR) of this combination therapy? What are the outcomes in terms of progression-free survival (PFS), overall survival (OS), and disease control rate (DCR)? What are the safety profiles and tolerability of the treatment?

Participants will receive:

Aipalolitovorelizumab (QL1706) injection at a dose of 5mg/kg, administered intravenously on Day 1 of each 3-week treatment cycle.

Fruquintinib at a dose of 5mg per day, taken orally continuously for the first 2 weeks of each 3-week cycle, followed by 1 week of withdrawal.

The treatment will continue until disease progression as assessed by RECIST v1.1 criteria, occurrence of unacceptable toxicity, decision to withdraw by the doctor or patient, non-compliance, or discontinuation due to administrative reasons. Participants will be monitored throughout the trial period to evaluate the efficacy and safety of the treatment.

DETAILED DESCRIPTION:
The immunodominant population in this study refers to the following:

* PD-L1 CPS score ≥ 10 points, and positive for tumor-infiltrating CD8+ T cells;

  * TMB ≥ 10 Muts/mb, and positive for tumor-infiltrating CD8+ T cells; ③ Functional mutations in epigenetic genes such as ARID1A, KMT2A/B/C/D, TET1/2/3, etc., and positive for tumor-infiltrating CD8+ T cells; ④ Presence of positive tertiary lymphoid structures (TLS) in the tumor microenvironment.

ELIGIBILITY:
Inclusion Criteria:

1. Have a full understanding of this study and voluntarily sign the informed consent form;
2. Aged 18 - 75 years;
3. Patients must be pathologically confirmed as advanced, metastatic or recurrent microsatellite stable (MSS) colorectal cancer (detected by immunohistochemistry, PCR or NGS according to the detection standards of each institutional testing center);
4. The results of patients' genetic testing show no POLD1/POLE mutations;
5. At least one immune marker is positive:

   * PD-L1 CPS score ≥ 10 points, and positive for tumor-infiltrating CD8+ T cells;

     * TMB ≥ 10 Muts/mb, and positive for tumor-infiltrating CD8+ T cells; ③ Functional mutations in epigenetic genes such as ARID1A, KMT2A/B/C/D, TET1/2/3, etc., and positive for tumor-infiltrating CD8+ T cells; ④ Presence of positive tertiary lymphoid structures (TLS) in the tumor microenvironment;
6. Patients have previously received two or more treatment regimens for advanced or metastatic colorectal cancer, at least one of which includes fluorouracil; or patients have previously received one treatment regimen for advanced or metastatic colorectal cancer and cannot tolerate the second-line standard chemotherapy regimen;
7. ECOG performance status of 0 - 1, with no deterioration within 7 days;
8. Expected survival ≥ 3 months;
9. Organ function levels must meet the following requirements:

   * Sufficient bone marrow reserve: absolute neutrophil count ≥ 1.5×10⁹/L, platelet count ≥ 90×10⁹/L, hemoglobin ≥ 9 g/dL; no blood transfusion or use of blood products within 14 days;

     * Liver: plasma albumin ≥ 2.8 g/dL; bilirubin ≤ 1.5 times the upper limit of normal (ULN); ALT and AST ≤ 2.5×ULN, and if there is liver metastasis, ALT and AST ≤ 5×ULN; ③ Kidney: serum creatinine ≤ 1.5×ULN;

       * Heart: left ventricular ejection fraction (LVEF) ≥ 50%; ⑤ Coagulation: prothrombin time (PT) ≤ 1.5×ULN, international normalized ratio (INR) ≤ 1.5×ULN, activated partial thromboplastin time (APTT) ≤ 1.5×ULN; ⑥ Thyroid-stimulating hormone (TSH) ≤ ULN (if abnormal, FT3 and FT4 levels should be examined simultaneously; if FT3 and FT4 levels are normal, patients can be enrolled);
10. Women of childbearing age need to take effective contraceptive measures;
11. Have good compliance and be cooperative with follow-up;
12. Agree to provide sufficient previously stored tumor tissue samples for testing.

Exclusion Criteria:

1. Unable to comply with the study protocol or research procedures;
2. Pregnant or lactating women;
3. Any factors affecting oral administration;
4. Patients who have previously received immunotherapy and fruquintinib;
5. Complicated with any of the following conditions: uncontrolled hypertension, coronary artery disease, arrhythmia, and heart failure;
6. Patients who participated in clinical studies of other drugs within 4 weeks before enrollment;
7. Alcohol or drug abuse within 4 weeks after the last clinical trial;
8. Anti-infective treatment did not stop 14 days before the start of the study;
9. Severe uncontrolled systemic diseases, such as severe active infections;
10. Urinalysis shows urine protein > ++, and it is confirmed that 24-hour urine protein > 1.0 g;
11. Active bleeding within 3 months; severe arterial/venous thrombotic events within 6 months; hereditary or acquired bleeding (e.g., coagulation dysfunction); major surgery (except biopsy and electroresection of polyps) within 4 weeks before the study, incompletely healed surgical incisions, or major trauma; use of aspirin (> 325 mg/day) or current or recent use of dipyridamole, clopidogrel, and cilostazol (10 days before the study);
12. Acute myocardial infarction, acute coronary syndrome, or coronary artery bypass grafting within 6 months before the first treatment;
13. Use of systemic glucocorticoids or other systemic immunosuppressive drugs within 2 weeks before treatment. Immunosuppressive drugs have been started or are expected to be used during the trial. Physiological replacement doses are allowed for inhaled glucocorticoids;
14. Fractures or long-term unhealed wounds;
15. Inactivated vaccines 接种 within 4 weeks before enrollment;
16. Having other malignant tumors within 5 years before enrollment, except for basal cell carcinoma or squamous cell carcinoma of the skin after radical resection, or carcinoma in situ of the cervix;
17. Known to be infected with human immunodeficiency virus (HIV), or positive for syphilis test, or known to be HIV-positive patients;
18. Previously received allogeneic bone marrow transplantation or organ transplantation;
19. Subjects allergic to the study drug or any of its auxiliary preparations;
20. Electrolyte abnormalities judged by the researcher to be clinically significant;
21. Detectable untreated chronic hepatitis B, chronic hepatitis B virus (HBV) carriers (HBV DNA > 2000 IU/mL), or HCV carriers with detectable HCV RNA. Note: Inactive hepatitis B surface antigen (HBsAg) carriers, treated and stable hepatitis B patients (HBV DNA < 2000 IU/mL) can be included in the study;
22. Previous radiation pneumonitis or chest CT scan showing active pneumonia within 4 weeks before the study;
23. The patient has an autoimmune disease requiring intervention;
24. Accompanied by brain metastasis, or severe malignant pleural or peritoneal effusion;
25. Any other diseases, clinically significant metabolic abnormalities, abnormal physical examination or laboratory test results, which, in the researcher's judgment, reasonably suggest that the patient has a disease or condition unsuitable for the use of the study drug (such as having epileptic seizures requiring treatment), or will affect the interpretation of study results, or put the patient at high risk;
26. Patients deemed inappropriate for inclusion in this study by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 6 months
  Objective Response Rate (ORR) refers to the proportion of patients who achieve complete response (CR) and partial response (PR) after treatment among the total number of evaluable patients.

SECONDARY OUTCOMES:
Progression Free Survival | 1 year
  Progression-Free Survival (PFS) refers to the time from the start of receiving treatment to the occurrence of objective tumor progression or the patient's death.
Overall survival | 2 years
  Overall survival defined as the time between signing the informed consent form to death due to various causes
Disease Control Rate | 6 months
  Disease Control Rate defined as the proportion of patients who achieved complete response (CR), partialresponse (PR), and stable disease (SD) according to RECIST v1.1.
Safety | 6 months
  Use NCl-CTCAE version 5.0 for classification and grading

CONTACTS AND LOCATIONS:
Overall Officials: Yanqiao Zhang, Principal Investigator — Harbin Medical University Cancer Hosptital